CLINICAL TRIAL: NCT04266834
Title: Establishing Clinical Utility of a New Diagnostic Test in Patients Undergoing Cardiac Catheterization: A CPV® Randomized Controlled Trial
Brief Title: Establishing Clinical Utility of a New Diagnostic Test in Patients Undergoing Cardiac Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qure Healthcare, LLC (Industry)
Collaborators: Hikari DX (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 01CMC2019
Record Dates: First submitted 2020-02-07; First posted 2020-02-12 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: AKI; Contrast-induced Nephropathy

STUDY DESIGN:
Intervention Model Description: The study will enroll practicing cardiologists in the US. All eligible and consented participants will be randomly assigned to either a control or intervention arm. All participants complete two rounds of three patient simulations. The intervention arm only will receive educational material about the Hikari L-FABP test in between these two rounds, and be provided simulated L-FABP test results in the second round of the simulated cases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Experimental-arm providers will complete two rounds of three simulated patient cases (CPVs) with two additions described in the next column:
  Interventions: Other: Experimental Arm
- Control (No Intervention): These providers will complete two rounds of three simulated patient cases (CPVs) only.

INTERVENTIONS:
Other: Experimental Arm — First, these providers will receive educational materials (e.g. a slide deck and one-page fact sheet) meant to mimic what physicians will receive in the real-world market as they learn about the Hikari DX L-FABP test.
  Second, within each of their second-round cases, intervention-arm physicians only will receive simulated test results from the L-FABP test at the clinically-appropriate point in each case.
  Arms: Experimental

SUMMARY:
This study will collect high-quality randomized controlled data across the U.S. from practicing cardiologists performing invasive/interventional procedures and determine how they currently manage patients at risk for CIN and how the results of Hikari's L-FABP test change clinical decision making.

DETAILED DESCRIPTION:
This study will collect high-quality randomized controlled data across the U.S. from practicing cardiologists performing invasive/interventional procedures and determine how they currently manage patients at risk for CIN and how the results of Hikari's L-FABP test change clinical decision making. Data from this study will better illuminate the clinical use cases with the most significant impact on clinical decision making (and thus the largest potential clinical utility) and the associated physician characteristics (e.g., age, practice setting, training) associated with test adoption.

This study leverages simulated patient cases called Clinical Performance and Value vignettes (CPVs) in a proven methodology to rapidly measure physician care decisions. CPVs are a unique and scalable tool that standardizes practice measurement by having all providers care for the same (virtual) patients. With all providers caring for the same patients, the CPVs generate unbiased data that yields powerful insights into clinical decision making and how these decisions change with the introduction of a new product or solution. Data from the CPVs can quickly demonstrate the clinical utility of a solution, be published in peer-reviewed literature, inform marketing strategies and positively impact coverage and reimbursement decisions.

The study is a prospective cohort trial with six steps:

1. Enrollment: The study will enroll 166 practicing cardiologists who perform invasive or interventional procedures in the U.S. and are determined to be eligible by an eligibility screener.
2. Provider survey: Once providers are enrolled in the study, they will be asked to complete a questionnaire describing their practice and professional background.
3. Randomization: The 166 cardiologists will be randomized into equally-sized (83) control and intervention arms.
4. CPVs (First Round): Physicians will complete three randomly-assigned CPV patient simulations in random order. Cases will be identical across the intervention and control arms. All cases are presented on an online platform, participants are provided with unique weblinks, accessible via any internet-connected computer.
5. Education: The intervention-arm cardiologists will receive educational materials duplicating what physicians would receive in the real-world market as they adopt the L-FABP test. These materials may be comprised of a slide deck, fact sheet, webinar, or case studies.
6. CPVs: Physicians will then complete three additional CPV patient simulations in random order. Cases will be identical across the intervention and control arms, except that the intervention arm will receive L-FABP test results at an appropriate point in each simulated case in the post-intervention round.

ELIGIBILITY:
Inclusion Criteria:

1. Board-certified in cardiology for at least two years
2. Averaging at least 20 hours per week of clinical and patient care duties over the last six months
3. Averaging at least one day per month performing invasive or interventional cardiology procedures over the last six months
4. English speaking
5. Access to the internet
6. Informed, signed and voluntarily consented to be in the study

Exclusion Criteria:

1. Non-English speaking
2. Unable to access the internet
3. Do not voluntarily consent to be in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
CPV-measured pre-/post-difference in quality scores between intervention and control physicians | 2-4 weeks
  All physicians' completed simulated CPV cases are scored based upon the quality of care provided. This measure CPV-measured pre-/post-difference in these care quality scores between control physicians using standard of care diagnostic tools and intervention physicians with access to L-FABP test results, including by use case types.
CPV-measured cost difference | 2-4 weeks
  Difference in expected cost of care between control and intervention physicians. (Cost will be calculated by measuring differential rates of medical interventions/levels of care selected by each arm, including by each use case, and multiplying by Medicare reimbursement rates for these interventions/levels of care, and/or by modeling the incidence of complications and calculating associated costs per above.)

SECONDARY OUTCOMES:
Baseline variation in CPV-measured quality scores | 1 week
  All physicians' completed simulated CPV cases are scored based upon the quality of care provided. This measure assesses the baseline levels of care quality variation in the work-up and management of patients at risk for CIN, including by use case types.

CONTACTS AND LOCATIONS:
Overall Officials: John Peabody, MD, PhD, Principal Investigator — President, QURE Healthcare
Locations (1):
- QURE Healthcare, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burgon TB, Cox-Chapman J, Czarnecki C, Kropp R, Guerriere R, Paculdo D, Peabody JW. Engaging Primary Care Providers to Reduce Unwanted Clinical Variation and Support ACO Cost and Quality Goals: A Unique Provider-Payer Collaboration. Popul Health Manag. 2019 Aug;22(4):321-329. doi: 10.1089/pop.2018.0111. Epub 2018 Oct 17. PMID 30328782
- [Background] Peabody JW, Strand V, Shimkhada R, Lee R, Chernoff D. Impact of rheumatoid arthritis disease activity test on clinical practice. PLoS One. 2013 May 7;8(5):e63215. doi: 10.1371/journal.pone.0063215. Print 2013. PMID 23667587
- [Background] Solon O, Woo K, Quimbo SA, Shimkhada R, Florentino J, Peabody JW. A novel method for measuring health care system performance: experience from QIDS in the Philippines. Health Policy Plan. 2009 May;24(3):167-74. doi: 10.1093/heapol/czp003. Epub 2009 Feb 18. PMID 19224955
- [Background] Peabody J, Martin M, DeMaria L, Florentino J, Paculdo D, Paul M, Vanzo R, Wassman ER, Burgon T. Clinical Utility of a Comprehensive, Whole Genome CMA Testing Platform in Pediatrics: A Prospective Randomized Controlled Trial of Simulated Patients in Physician Practices. PLoS One. 2016 Dec 30;11(12):e0169064. doi: 10.1371/journal.pone.0169064. eCollection 2016. PMID 28036350
- [Background] Peabody JW, Luck J, Glassman P, Jain S, Hansen J, Spell M, Lee M. Measuring the quality of physician practice by using clinical vignettes: a prospective validation study. Ann Intern Med. 2004 Nov 16;141(10):771-80. doi: 10.7326/0003-4819-141-10-200411160-00008. PMID 15545677